CLINICAL TRIAL: NCT04232059
Title: The Effect of Different Ventilation Strategies on Cerebral Oxygenation Using Near Infrared Spectroscopy (NIRS) in Pediatrics Undergoing Posterior Fossa Tumor Surgery: Randomized Controlled Cross Over Study
Brief Title: The Effect of Different Ventilation Strategies on Cerebral Oxygenation Using Near Infrared Spectroscopy (NIRS) in Pediatrics Undergoing Posterior Fossa Tumor Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kasr El Aini Hospital (Other)
Responsible Party: Principal Investigator, Khaled Abdelfattah Abdallah Sarhan, lecturer of anesthesia, Kasr El Aini Hospital
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Diagnostic
Other Study IDs: MD-X-2020
Record Dates: First submitted 2020-01-12; First posted 2020-01-18 (Actual); Last update posted 2022-03-07 (Actual); Status verified 2021-03

CONDITIONS: Infratentorial Neoplasms; Hyperventilation; Craniotomy
Keywords: posterior fossa; cerebral oximetry; hyperventilation; children
MeSH Terms: conditions — Infratentorial Neoplasms; Hyperventilation

STUDY DESIGN:
Intervention Model Description: The aim of this study is to evaluate the changes of cerebral oxygen saturation during hyperventilation and normo-ventilation (using near-infrared spectroscopy) in pediatrics undergoing posterior fossa tumor resection.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1: hyperventilation (Active Comparator): • Group 1: hyperventilation (ETco2 25-30 mm Hg) for 20 minutes that will start immediately after skin incision followed by normoventilation (ETco2 31-35 mm Hg) for another 20 minutes.
  Interventions: Device: cerebral oximetry
- Group 2: normoventilation (Active Comparator): • Group 2: normoventilation (ETco2 31-35 mm Hg) for 20 minutes immediately after skin incision followed by hyperventilation (ETco2 25-30 mm Hg) for another 20 minutes.
  Interventions: Device: cerebral oximetry

INTERVENTIONS:
Device: cerebral oximetry — evaluation of the changes of cerebral oxygen saturation during hyperventilation and normo-ventilation (using near-infrared spectroscopy) in pediatrics undergoing posterior fossa tumor resection.

SUMMARY:
The aim of this study is to evaluate the changes of cerebral oxygen saturation during hyperventilation and normo-ventilation (using near-infrared spectroscopy) in pediatrics undergoing posterior fossa tumor resection.

DETAILED DESCRIPTION:
Introduction:

Hyperventilation has been used for intraoperative brain relaxation for decades, Interestingly, this common practice is not based on robust evidence .

The mechanism of brain relaxation secondary to hyperventilation is attributed to the hypocapnia induced cerebral vasoconstriction and the subsequent reduction of cerebral blood volume (CBV) and intracranial volume. The CBV reduction is accompanied by the reduction in cerebral blood flow that could render the brain at ischemic risk, if the cerebral metabolic activity remains the same before and after hyperventilation. So, it is possible that inadvertent cerebral ischemia may outweigh the benefits of hyperventilation and should be subjected for further investigation.

Cerebral near-infrared spectroscopy (NIRS) is a useful non-invasive tool for regional cerebral oxygen saturation (rScO2) monitoring, which provides continuous, real time information on the balance between cerebral oxygen delivery and consumption.

Cerebral oximetry monitoring had the ability to detect clinically silent episodes of cerebral ischemia in a variety of clinical settings which could be an important safeguard for cerebral function.

Hyperventilation had been shown to significantly reduce cerebral oxygenation using near-infrared spectroscopy in patients undergoing elective abdominal surgery.

Multiple studies have shown that prolonged hyperventilation correlated with poor outcome especially in brain injured patients. 5,6 However, there is still a lack of evidence on the relationship between hyperventilation and neurological outcome in patients having craniotomy.

However, to the best of the investigator's knowledge no previous randomized controlled trials had studied the effect of hyperventilation versus normo-ventilation on cerebral oximetry in pediatrics undergoing posterior fossa tumor surgeries.

V. Study procedure:

This is a prospective, randomized controlled trial with a two-period crossover design so that the patient can act as a control to himself. Enrolled patients are children (1-6 years old) undergoing posterior fossa tumor resection. Prior to anesthetic induction, the two sensors (SAFB-SM, Covidien, Dublin, Ireland) for near-infrared spectroscopy (INVOS 5100C, Covidien, Dublin, Ireland) will be applied on the left and right sides of the forehead with the caudal border approximately 1 cm above the eyebrows to measure regional oxygen saturation (rSO2). A bispectral index (BIS) sensor will also be fixed on the left forehead (Model QUATRO, Covidien, Dublin, Ireland) to monitor the depth of anesthesia. Both sensors will be fixed to their positions using adhesive pads to avoid removal during positioning and soaking with betadine solution. Baseline values for cerebral oxygen saturation will be obtained using NIRS monitor, Standard monitors (electrocardiogram, non-invasive blood pressure, pulse oximeter) will be applied to all patients. The anesthetic management will be standardized for all patients as follows:

General anesthesia will be induced by inhalational agent 'sevoflurane' until intravenous line is secured then Fentanyl (1-2 µg/kg), Propofol (1-2 mg/Kg) will be given intravenously. Intubation will be facilitated by Atracurium (0.5 mg/kg) and confirmed by capnography. Nasopharyngeal temperature probe will be inserted for monitoring of core body temperature which will be kept between 36.5-37 C using warming blankets. A 22 G arterial cannula will be placed in the left radial artery and baseline ABG will be obtained to correlate value of Etco2 and Paco2. Anesthesia will be maintained with isoflurane in oxygen 40% and will be adjusted to maintain BIS between 40 and 60 and Atracurium infusion (0.5 mg/kg/hr). Central venous line will be inserted in the right internal jugular vein under complete aseptic condition under ultrasound guidance, wide bore peripheral cannula will be inserted for fluid management and a Foley's catheter will be inserted in the urinary bladder for urine output monitoring. Patients will be positioned in the prone position with the arms positioned and secured at the patient's side and after careful padding of the pressure points; the patient head will be supported on the forehead using a horseshoe adapter. Slight neck flection will be permitted till the anesthetist can pass two fingers easily between the chin and the chest to allow for optimum surgical exposure. Patients will be randomly assigned using concealed envelopes, according to a computer-generated random number to one of the following two treatment sequences:

* Group 1: hyperventilation (ETco2 25-30 mm Hg) for 20 minutes that will start immediately after skin incision followed by normoventilation (ETco2 31-35 mm Hg) for another 20 minutes.
* Group 2: normoventilation (ETco2 31-35 mm Hg) for 20 minutes immediately after skin incision followed by hyperventilation (ETco2 25-30 mm Hg) for another 20 minutes. The ventilation strategies will be achieved using volume-controlled mode with a tidal volume of 8 ml/kg, I/E ratio:1/2 and ETco2 will be maintained at the desired range by adjusting the respiratory rate. Positive end-expiratory pressure (PEEP) will not be applied. After removal of the bone flap and exposure of the dura matter, a 20-gauge plastic cannula will be inserted into the subdural space along the surface of the brain. This will be connected to a calibrated pressure transducer via a length of polyethylene high pressure tubing filled with normal saline. The transducer will be zeroed at ear level. During the study period, the mean subdural pressure will be recorded at 2 minutes intervals at the end expiratory phase.

Assessment phase 1: An arterial blood sample will be obtained immediately after skin incision for blood gas analysis to determine the difference between arterial and end-tidal carbon dioxide tension (Pa-ETCO2). Ventilation and ETCO2 will be kept constant for at least 20 min, which is long enough for stabilization of any vascular responses to the change in Paco2. At the end of the equilibration period (20 minutes), another arterial blood sample will be obtained to confirm that the targeted Paco2 (was achieved. The neurosurgeon, unaware of the anesthetic and ventilatory management provided, will be then asked to score the brain bulk according to a four-point scale as follows:

1. Excellent with no swelling
2. Minimal swelling, acceptable
3. Swollen but no treatment required
4. Swollen, needing treatment. After this assessment, ventilation will be changed immediately according to group assignment.

Assessment phase 2: Another 20 min of equilibration will be allowed and measurements will be repeated as previously described. During the whole period of study (40 minutes), the cerebral oximetry will be recorded at 5 minutes intervals. During this period factors that may affect cerebral oximeter will be controlled by maintaining position of the patient head, (normothermia with temperature at 36.5-37 C), within 20% of the base line blood pressure using increments of ringer solution and ephedrine boluses as appropriate, maintain PH 7.35-7.45, Hb level around 10 gm/dl guided by blood loss and repeated measurements of Hb in ABG and blood glucose level between 80-180 mg/dl. The study will be ended at this point, the subdural cannula will be removed, and surgery will proceed as normal. Specific or routine interventions for brain swelling such as a change in body position or diuretic therapy with mannitol or furosemide will not be administered until the study had ended. However, for ethical reasons, interventions will be made if requested by the surgeon and the patient will be then withdrawn from the study. Data will be collected by an independent blinded anesthesiologist using a data collection form.

• Measurement tools:

* Demographic and categorical characteristics including patient's age in years, weight in Kg, gender, type of the procedure( 4th ventricular, medulloblastoma,... )
* Both NIRS values at baseline and every 5 minutes during each phase of the study
* Subdural intracranial pressure (ICP) every 2 minutes during each phase of the study
* End tidal co2 every 5 minutes during each phase of the study
* Paco2 baseline and at the end of each phase of ventilation (20 minutes following start of phase 1 assessment and 20 minutes after start of phase 2 assessment)
* Heart rate and mean arterial blood pressure every 10 minutes.
* Brain relaxation score

ELIGIBILITY:
Inclusion Criteria:

- Age : 1 to 6 years old

* Both sexes
* ASA I-II
* scheduled for posterior fossa tumor resection.

Exclusion Criteria:

* Age < 1 year or > 6 years old

  * Comorbid condition (ASA classification > II)
  * patient with anemia (Hb <10 g/dl)
  * Emergency surgery
  * Patients with VP shunt, on diuretics, recurrent tumors, cerebral infarction and or hemorrhage
  * Patients on cardiovascular support e.g.:, inotrope or vasoconstrictor infusions

Ages: 1 Year to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 42 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2021-12-01 (Actual); Study Completion 2021-12-01 (Actual)

PRIMARY OUTCOMES:
NIRS value at the end of phase 1 assessment in each group | 20 minutes after skin incision
  NIRS value at the end of phase 1 assessment in each group

SECONDARY OUTCOMES:
- Brain relaxation score | 20 minutes after skin incision
  Brain relaxation score: four-point scale as follows:
  1. Excellent with no swelling
  2. Minimal swelling, acceptable
  3. Swollen but no treatment required
  4. Swollen, needing treatment. the higher the score the higher the intracranial pressure
- Subdural intracranial pressure (ICP) | Subdural ICP every 2 minutes during each phase of the study (40 minutes)
  - Subdural intracranial pressure (ICP)

CONTACTS AND LOCATIONS:
Locations (1):
- Kasralainy, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided